CLINICAL TRIAL: NCT02630160
Title: The Influence of Local Infiltration Analgesia by Catheter in Postoperative Control Pain After Total Hip Replacement
Acronym: ILIACPCPTHR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Daniel Pérez Prieto, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/5138/I
Record Dates: First submitted 2015-11-30; First posted 2015-12-15 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2015-12

CONDITIONS: Musculoskeletal Pain; Hip Injuries
MeSH Terms: conditions — Musculoskeletal Pain; Hip Injuries | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intraarticular Catheter with anesthesic (Active Comparator): Intraarticular infusion with Bupivacaine Hydrochloride
  Interventions: Drug: Bupivacaine hydrochloride
- Intraarticular Physiological Saline (Placebo Comparator): Infusion of Physiological Saline [Flebobag Salina Fisiologica Grifols 0.9%] Sterile Solution by intraarticular catheter
  Interventions: Other: Physiological Saline
- Perifascial Catheter with anesthesic (Active Comparator): Perifascial infusion with Bupivacaine Hydrochloride
  Interventions: Drug: Bupivacaine hydrochloride
- Perifascial Physiological Saline (Placebo Comparator): Infusion of Physiological Saline [Flebobag Salina Fisiologica Grifols 0.9%] Sterile Solution by Perifascial catheter
  Interventions: Other: Physiological Saline

INTERVENTIONS:
Drug: Bupivacaine hydrochloride — Intraarticular infusion with bupivacaine
  Other Names: Bupivacaine / epinephrine, Vivacaine
  Arms: Intraarticular Catheter with anesthesic; Perifascial Catheter with anesthesic
Other: Physiological Saline — Intraarticular infusion physiological serum
  Other Names: Flebobag Salina Fisiologica Grifols 0.9%
  Arms: Intraarticular Physiological Saline; Perifascial Physiological Saline

SUMMARY:
A randomized double-blind clinical trial was performed. There were 4 groups according to catheter placement and infusion constituents: 1) Intraarticular catheter + anesthetics; 2) Intraarticular catheter +placebo; 3) Subfascial catheter + anesthetics; 4) Subfascial catheter + placebo. The anesthetics infusion contained bupivacaine (bolus + continuous perfusion up to 36 hours). The placebo solution consisted in physiological serum (bolus + continuous perfusion up to 36 hours). Randomization was performed in the hospital pharmacy and the surgeon kept out the surgical field when the resident placed the catheter. The same conventional analgesic schedule was prescribed to all patients: PCA (patient controlled analgesia) + paracetamol 1g/6h + dexketoprofen 50mg/12h. The pain was evaluated by means of PCA (patient controlled analgesia) shots and the VAS (visual analog scale). Side effects, time to start rehabilitation and time to discharge were also analyzed. A statistical analysis was performed to compare all this variables between the 4 groups (SPSS 18.0).

ELIGIBILITY:
Inclusion Criteria:

* Primary total Hip Replacement

Exclusion Criteria:

* Allergic to Bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in pain measured with a visual analog scale | 36 hours
  Visual analog pain scale score every eight hours for 36 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pérez Prieto, Principal Investigator — Hospital del Mar; Marta Cuenca Llavall, Study Chair — Hospital del Mar; Fernando Marques Lopez, Study Director — Hospital del Mar; Alfonso Leon Garcia, Study Chair — Hospital del Mar; Francisco Javier Santiveri Papiol, Study Chair — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain